CLINICAL TRIAL: NCT05825664
Title: Comparison of the Efficiency and Safety of Underwater Endoscopic Mucosal Resection and Conventional Endoscopic Mucosal Resection in the Treatment of Non-pedunculated Colorectal Polyps
Brief Title: Underwater Versus Conventional Endoscopic Mucosal Resection in the Treatment of Non-pedunculated Colorectal Polyps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Le Dinh Quang, Principal investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2023-04-07; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Colorectal Polyp; Colorectal Neoplasms
Keywords: colorectal polyp; underwater endoscopic mucosal resection; conventional endoscopic mucosal resection
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Underwater endoscopic mucosal resection (Experimental): Intervention: Non-pedunculated polyps will be removed by underwater endoscopic mucosal resection. The UEMR procedure included the following: (1) complete deflation of the colorectal lumen; (2) total immersion of the lesion in normal saline using a mechanical water pump; (3) snaring the lesion and the surrounding mucosa; and (4) resection using electrocautery.
  Interventions: Procedure: Endoscopic resection
- Conventional endoscopic mucosal resection (Active Comparator): Intervention: Non-pedunculated polyps will be removed by conventional endoscopic mucosal resection. The CEMR procedure included the following: (1) needle injection of normal saline into the submucosa; (2) entrapment of the mucosal protrusion with a snare; and (3) resection applying the same electrocautery setting as was used for UEMR.
  Interventions: Procedure: Endoscopic resection

INTERVENTIONS:
Procedure: Endoscopic resection — Group 1: Polyps are resected by UEMR Group 2: Polyps are resected by CEMR

SUMMARY:
A prospective, randomized, controlled study to compare the efficacy and safety of underwater endoscopic mucosal resection and conventional endoscopic mucosal resection in removal of non-pedunculated colorectal polyps

DETAILED DESCRIPTION:
* Patients are undergone colonoscopy at the Endoscopy department of Ho Chi Minh City University Medical Center.
* Randomize patients with non-pedunculated polyp of 10mm or larger in size into 2 interventional groups based on Random function of Statistical Package for the Social Sciences (SPSS) 20.0, including (1) Group 1: Underwater endoscopic mucosal resection (UEMR) and (2) Group 2: Conventional endoscopic mucosal resection (CEMR).
* The time of local recurrence assessment depends on the histopathology of polyps. Polyps with low grade dysplasia are followed up at 6 months, while polyps with high grade dysplasia are followed at 3 months.
* Collecting variables which consist of primary and secodary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Non-pedunculated polyps of 10 mm or more in size
* Type 1 or 2 according to NBI International Colorectal Endoscopy (NICE) classification
* Patients must sign an informed consent form prior to registration in study

Exclusion Criteria:

* Lesions with signs of deep invasion (hard, friable tissue, poor mobility, positive "non-lifting" sign)
* Type 3 according to NICE classification
* Colorectal cancer
* Patients with unstable chronic disease (melitus diabetes, hypertension, heart failure, kidney failure, liver failure, chronic obstructive pulmonary disease)
* Hemostasis disorder (INR > 1.5; platelets < 100000/mm3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2023-04-07 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
en bloc resection | immediately after the procedure
  Rate of en bloc resection for non-pedunculated colorectal polyps of 10 mm or more
Curative rate | through study completion, an average of 6 months
  Curative rate for non-pedunculated colorectal polyps of 10 mm or more

SECONDARY OUTCOMES:
Complication rate | up to 2 weeks
  Rate of complications including bleeding, perforation
Local recurrence rate | 6 months
  Rate of local recurrence
Procedure time | during the procedure
  Time for complete resection of polyps

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medicine and Pharmacy at Ho Chi Minh city, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No